CLINICAL TRIAL: NCT05009940
Title: A Clinical Investigation Evaluating the Efficacy of Gradusox™ Compression Hosiery at Enhancing Dermal Oxygen Levels in Healthy Participants Post-varicose Vein Surgery.
Brief Title: Skin Oxygenation Whilst Wearing Gradusox™ Compression Hosiery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Whiteley Clinic (Other)
Collaborators: VeinSense (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TWC-AC-2021-02
Record Dates: First submitted 2021-08-13; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Effect of Compression Hosiery on the Local Tissue Oxygenation and Compare This Effect Against That Achieved by Standard Compression Hosiery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gradusox then Sigvaris compression stockings (Experimental): This arm refers to the order of interventions received by the participant. The first intervention received by participants in this arm are Gradusox compression stockings applied to both legs.
  After a washout period, the second intervention received are Sigvaris compression stockings applied to both legs.
  Interventions: Device: Graduated compression stockings
- Sigvaris then Gradusox compression stockings (Experimental): This arm refers to the order of interventions received by the participant. The first intervention received by participants in this arm are Sigvaris compression stockings applied to both legs.
  After a washout period, the second intervention received are Gradusox compression stockings applied to both legs.
  Interventions: Device: Graduated compression stockings

INTERVENTIONS:
Device: Graduated compression stockings — Both GraduSOX and Sigvaris are graduated compression stockings. These exert the greatest degree of of compression at the ankle, and the level of compression gradually decreases up the garment.
  Other Names: GraduSOX; Sigvaris

SUMMARY:
The primary objective is to evaluate the effect of Gradusox™ compression hosiery on the local tissue oxygenation and compare this effect against that achieved by standard compression hosiery.

DETAILED DESCRIPTION:
After being informed about the study, all participants giving written informed consent will be randomised by closed envelope randomisation to either a) first, GraduSOX on their right leg and Sigvaris on their left leg, then GraduSOX on their left leg and Sigvaris on their right leg, or b) first, GraduSOX on their left leg and Sigvaris on their right leg, then GraduSOX on their right leg and Sigvaris on their left leg.

Participants will attend the clinic and be fitted with their stockings. Non-invasive probes will be taped to the skin above the inner ankle on both legs - these take measurements for SO2, oxyHb and deoxyHb every second. Measurements for these variables will be taken for 15 minutes whilst participants are not wearing stockings, as well as with stockings (worn in the order assigned to them). During these 15 minutes, participants will lie in supine for 5 minutes, then in sitting position for 5 minutes, then will return to supine for the last 5 minutes.

Between each stocking, participants will be asked to take a 10 minute walk and return to the recliner in supine to re-equilibrate for a further 15 minutes.

The total time that measurements are taken for per participant is 50 minutes.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 and over.
* Have known previous venous insufficiency that has been treated.
* Have no known current contraindication to the wearing of graduated compression hosiery.
* Have an ankle brachial pressure index (ABPI) between 0.8-1.2.
* Have no active ulceration.
* Are physically able to apply and remove hosiery kits safely.
* Have had successful surgery at The Whiteley Clinic and have had at least one follow-up to show no residual venous disease.

Exclusion Criteria

* Under the age of 18.
* Have known arterial insufficiency (an ABPI of below 0.8).
* Have active ulceration.
* Be physically unable to put stocking on their own legs.
* Have signs of recent lower limb trauma, active infection, ongoing untreated venous disease, significant ankle oedema.
* Unable to give informed consent.
* Pregnant.
* Fragile skin that may be damaged whilst trying to apply or remove compression stockings.
* Previous DVT or complicated varicose veins that were not able to be completely treated and left residual venous reflux disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
SO2 | 50 minutes
  Transcutaneous oxygen saturation
OxyHb | 50 minutes
  Oxyhaemoglobin
DeoxyHb | 50 minutes
  Deoxyhaemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS FRCS(Gen) MBBS, Principal Investigator — The Whiteley Clinic
Locations (1):
- The Whiteley Clinic, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participants that are enrolled in the study will be assigned a unique Trial ID which will be used to anonymise data related to themselves.

REFERENCES:
- [Background] Nelson EA, Adderley U. Venous leg ulcers. BMJ Clin Evid. 2016 Jan 15;2016:1902. PMID 26771825
- [Background] Phillips CJ, Humphreys I, Thayer D, Elmessary M, Collins H, Roberts C, Naik G, Harding K. Cost of managing patients with venous leg ulcers. Int Wound J. 2020 Aug;17(4):1074-1082. doi: 10.1111/iwj.13366. Epub 2020 May 7. PMID 32383324
- [Background] Evans SR. Clinical trial structures. J Exp Stroke Transl Med. 2010 Feb 9;3(1):8-18. doi: 10.6030/1939-067x-3.1.8. PMID 21423788